CLINICAL TRIAL: NCT06282211
Title: A Multicenter, Open-label, Randomized Controlled Clinical Study of the Efficacy and Safety of Ondansetron Oral Soluble Pellicles for the Prevention of Delayed Nausea and Vomiting Induced by Highly Emetogenic Chemotherapy
Brief Title: the Efficacy and Safety of Ondansetron Oral Soluble Pellicles
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The First Affiliated Hospital of Xinxiang Medical College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHASE 005
Record Dates: First submitted 2023-12-19; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Nausea and Vomiting
MeSH Terms: conditions — Nausea; Vomiting

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ondansetron Oral Soluble Pellicles (Experimental): nausea and vomiting prophylaxis with Ondansetron Oral Soluble Pellicles, 8 mg tid for 5-7 days after chemotherapy
  Interventions: Drug: Ondansetron Oral Soluble Pellicles
- no antiemetic drugs or drugs with antiemetic active ingredients (Sham Comparator): no antiemetic drugs or drugs with antiemetic active ingredients for 5-7 days after chemotherapy
  Interventions: Drug: Ondansetron Oral Soluble Pellicles

INTERVENTIONS:
Drug: Ondansetron Oral Soluble Pellicles — patients applying cisplatin-based chemotherapy regimen were treated with the triple combination of fosaprepitant (Tanneng, Jiangsu Haosen Pharmaceutical Group Co., Ltd.) + Ondansetron Oral Soluble Pellicles (Aiqisu, Jiangsu Hengrui Pharmaceutical Co., Ltd.) + dexamethasone for the prophylaxis of nausea and vomiting prior to the chemotherapy, and were divided into the experimental group and the control group by whether or not to continue the prophylaxis with o Ondansetron Oral Soluble Pellicles for 5-7 days after the chemotherapy as shown in the figure below.
  Other Names: Aiqisu

SUMMARY:
The name of this prospective study is a multicenter, open-label, randomized controlled clinical study of the efficacy and safety of Ondansetron Oral Soluble Pellicles for the prevention of delayed nausea and vomiting induced by highly emetogenic chemotherapy.

DETAILED DESCRIPTION:
The aim of this study is to observe the efficacy and safety of ondansetron in delayed nausea and vomiting by its continuous dosing, and it is planned to enroll 184 first-time recipients of highly emetogenic single-day chemotherapy regimens (cisplatin dose 60-75 mg/m2; anthracycline compounds adriamycin ≥ 60 mg/m2 or epothilone ≥ 90 mg/m2 ) who were initiated on a triple combination regimen of fosaprepitant + ondansetron orally soluble film + dexamethasone triple regimen for nausea and vomiting prophylaxis in patients. The primary observation was the incidence and severity of delayed nausea and vomiting in both groups from day 5 after chemotherapy to the second cycle of chemotherapy. The secondary observation indexes include the incidence and severity of delayed nausea in patients in both groups from day 5 after chemotherapy to before the second cycle of chemotherapy; the incidence and severity of anticipatory nausea/vomiting in the second cycle of chemotherapy in both groups; the incidence and severity of nausea/vomiting in patients in both groups on days 1-4 after chemotherapy; and the incidence of adverse events and serious adverse reactions, with a focus on the antiemetic drugs common constipation, headache and other events. This trial was randomized into groups, and the experimental group was preset as group A and the control group as group B. The prevention of nausea and vomiting was carried out with the triple regimen of fosaprepitant (Tanneng, Jiangsu Hausen Pharmaceutical Group Co., Ltd.) + Ondansetron Oral Soluble Pellicles (Aiqisu, Jiangsu Hengrui Pharmaceutical Co., Ltd.) + dexamethasone prior to chemotherapy, and the patients were divided into the treatment group A and the control group B by the use of Ondansetron Oral Soluble Pellicles for continuation of the prophylaxis on the 5-7 days after the chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years, gender is not limited;
2. Histologically or cytologically confirmed diagnosis of malignant solid tumor;
3. Initial highly emetogenic one-day chemotherapy regimen (cisplatin dose 60-75 mg/m2; anthracycline compound adriamycin ≥ 60 mg/m2 or epothilone ≥ 90 mg/m2 ); and
4. Nausea and vomiting prophylaxis with a triple regimen of fosaprepitant + ondansetron orally dissolved membrane + dexamethasone started before chemotherapy;
5. Expected survival ≥ 3 months;
6. Eastern Cooperative Oncology Group (ECOG) physical status score ≤2;
7. Patients were able to read, understand, and complete study questionnaires;
8. Patients understood the study procedures and signed a written informed consent form

Exclusion Criteria:

1. Patients scheduled to receive multiple days of highly emetogenic chemotherapy within one week;
2. Patients using an antiemetic drug other than the study drug or a drug with an antiemetic active ingredient within 48 h prior to initiation of randomization and/or within one week of enrollment;
3. Symptoms such as vomiting prior to randomization;
4. Patients on opioid therapy (except stable dose administration);
5. Patients treated with a chemotherapy regimen containing generic paclitaxel (using castor oil as a solvent);
6. Patients who have received, or are expected to receive, radiotherapy to the abdomen (including the diaphragmatic plane and below) or pelvis within 1 week before randomization or one week after enrollment;
7. Patients with active infection (e.g., pneumonia) or any uncontrolled disease (e.g., diabetic ketoacidosis, gastrointestinal obstruction) other than malignancy;
8. The patient has participated in another clinical trial within the past 4 weeks;
9. Any condition that, in the judgment of the investigator, is unstable or may jeopardize the safety of the subject and his or her compliance with the study;
10. Pregnant or lactating females;
11. Presence of allergic conditions or prior serious adverse reactions to the study drug and excipients;
12. Suffering from psychological, familial, social, or geographic conditions that may prevent compliance with the study protocol and follow-up schedule;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2024-02-20 (Estimated); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-12-29 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of delayed vomiting in patients from day 5 after chemotherapy until the second cycle of chemotherapy in both groups | 21 days
  The incidence of delayed vomiting was recorded and the severity of delayed vomiting was assessed by the VAS scale.

SECONDARY OUTCOMES:
Incidence and severity of delayed nauseating in patients from day 5 after chemotherapy until the second cycle of chemotherapy in both groups | 21 days
  The incidence of delayed nauseating was recorded and the severity of delayed nauseating was assessed by the VAS scale.
Incidence and severity of nausea/vomiting in patients on days 1-4 after chemotherapy in both groups | 4 days
  The incidence of delayed nausea/vomiting was recorded and the severity of delayed nausea/vomiting was assessed by the VAS scale.

OTHER OUTCOMES:
Incidence of adverse events and serious adverse reactions throughout the study period | 21 days
  Record the incidence of adverse events and serious adverse reactions throughout the study period, focusing on events such as constipation and headache, which are common with antiemetics

CONTACTS AND LOCATIONS:
Locations (1):
- Keya Zhi, Weihui, None Selected, China

IPD SHARING:
Plan to Share IPD: No